CLINICAL TRIAL: NCT03872310
Title: A Study of Cognitive Enhancement of Transcranial Direct Current Stimulation on Working Memory in Patients With Schizophrenia
Brief Title: Cognitive Enhancement on Working Memory in Patients With Schizophrenia
Acronym: CEWMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Wang Jiunn-Kae, Attending physician of psychiatry department, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: N201701040
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Memory Deficits; Schizophrenia; Neurostimulator; Complications
Keywords: Schizephrenia; Cognitive enhancement; Transcranial direct current stimulation; Non-invasive brain stimulation; Working memory
MeSH Terms: conditions — Memory Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active comparator (Active Comparator): Within group
  Interventions: Device: STARSTIM
- Sham comparator (Sham Comparator): Within group
  Interventions: Device: STARSTIM

INTERVENTIONS:
Device: STARSTIM — Right DLPC was located as F4 according to the international 10-20 EEG system. Anodal tDCS was delivered with the anodal pole on the right DLPFCand the cathodal pole on the left cheek of the participant to avoid contaminating other brain regions during electrical stimulation via a pair of rubber electrodes housed in saline-soaked sponge coverings (5x5 cm^2). The direct current was applied with 1.5 mA for 15 min which can facilitate visual short-term memory and create an excitatory effect for up to 90 min. The anodal tDCS stimulated the right DLPC for 15 min with 1.5 mA in active tDCS condition. The sham tDCS condition followed identical tDCS protocol and same 15-min duration except the stimulation time only lasted for the initial 30s so that the participants felt the same initial tingling sensation (if any, only in some participants) but without the actual stimulation. The investigators will perform assessments of adverse effects after each session by a standardized questionnaire.

SUMMARY:
The investigators plan to investigate the effect of enhancement on working memory (WM) in patients of chronic schizophrenia and determine the predictive factors of effective treatment.

DETAILED DESCRIPTION:
Schizophrenia is a chronic and disabling disease with a prevalence of 0.5%~1.5% in the general population. It's estimated 98% of patients with schizophrenia exhibit variable degrees of cognitive deficits which have been well established to be predictive of patient functioning. A number of treatments had been developed for cognitive enhancement in patients with schizophrenia, nevertheless none of them showed satisfying results.

Transcranial direct current stimulation (tDCS) is a safe and convenient treatment which has showed some evidence of beneficial effects on working memory (WM) in both healthy and neuropsychiatric populations. However, studies of tDCS for cognitive enhancement in patients with schizophrenia are still quiet limited. The results of our previous studies in healthy participants and patients with diabetic polyneuropathy suggest that the anodal tDCS over right dorsolateral prefrontal cortex (DLPFC) improved spatial WM capacity, particularly when task difficulty demands more complex mental manipulations and for the low-performing patients in baseline assessments. Thus, we hypothesize that in the baseline the more severe the patients' cognitive deficit are, the greater their WM capacity improvement would be after applying the anodal Tdcs over right DLPFC.

The investigators plan to recruit 40 patients with chronic schizophrenia. First, the investigators will collect baseline characteristics including disease severity, cognitive deficits and brain connectivity. Then the investigators will adopt a sham-active crossover design for tDCS treatment with the order of the two sessions (sham and active) counterbalanced across participants. The investigators will perform pre- tDCS and post- tDCS assessments of their spatial WM and verbal WM as well as statistical analyses to see if the effect of cognitive enhancement reaches a significant level. In addition, the investigators will explore the possible predictive indicators of effective treatment.

ELIGIBILITY:
Inclusion criteria

1. Inform consent acquired
2. Age 20 to 50
3. Right-handed
4. Patients with schizophrenia diagnosed according to DSM-5 criteria

Exclusion criteria

1. Participants who are pregnant or breastfeeding
2. Participants who have metal implants
3. Participants who have alcohol/substance use disorder or received electro-convulsive therapy within the past 6 months.
4. Participants who have history of head injury with loss of consciousness
5. Participants who have history of brain lesions, infection, or epilepsy
6. Skin lesions on the electrodes placed
7. Cancer patients
8. Patients with high fever
9. Patients with significant sensory loss

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Visual-spatial working memory span measured by Corsi Block-Tapping task | up to one hour
  The paradigm was computer-adaptive, and thus the set size would only increase if the participant passed consecutive two trials of the same span. The lowest span level started from 2 (2 squares that change color) and up to 9 as maximum.
Verbal working memory measured by digit-span test | up to one hour
  The paradigm was also computer-adaptive

CONTACTS AND LOCATIONS:
Overall Officials: Jiunn-Kae Wang, MD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Shuang-Ho Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No